CLINICAL TRIAL: NCT04472676
Title: A Safety, Tolerability, and Pharmacokinetic Study of Single-and Multiple-Ascending Doses of LY3473329 in Healthy Subjects
Brief Title: A Study of LY3473329 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17611; J2O-MC-EKBA (Other: Eli Lilly and Company); 2020-002522-91 (EudraCT Number)
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3473329 (Part A) (Experimental): LY3473329 administered orally.
  Interventions: Drug: LY3473329
- Placebo (Part A) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- LY3473329 (Part B) (Experimental): LY3473329 administered orally.
  Interventions: Drug: LY3473329
- Placebo (Part B) (Experimental): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3473329 — Administered orally.
  Arms: LY3473329 (Part A); LY3473329 (Part B)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study in healthy participants is to learn more about the safety of LY3473329 and any side effects that might be associated with it. Blood tests will be performed to check how much LY3473329 gets into the bloodstream and how long the body takes to eliminate it. This is a two-part study. Participants may only enroll in one part.

For each participant:

* Part A will last up to about 19 weeks and may include 9 visits.
* Part B will last up to about 28 weeks and may include 11 visits.

ELIGIBILITY:
Inclusion Criteria:

* Males and females must adhere to contraception restrictions
* Have clinical laboratory test results within normal reference range or with acceptable deviations
* Body mass index (BMI) less than or equal to (≤)30 kilograms per square meter (kg/m²)
* For Part B:

  * Lipoprotein (a) (Lp[a]) greater than or equal to (≥)75 nanomoles per Liter (nmol/L) or 30 milligrams per deciliter (mg/dL) at screening
  * Plasminogen is within the normal range at screening

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the past 30 days from, a clinical trial involving an investigational drug that has not received regulatory approval for any indication, except for any trial involving antisense Lp(a), for which 6 months must have passed from the participant's last study drug dose
* Have previously completed or withdrawn from this study or any other study investigating LY3473329
* Are pregnant or breast feeding
* Glomerular filtration rate (GFR) is lower than estimated GFR 60 milliliters per minute per 1.73 square meters (mL/min/1.73 m2) using the Modification of Diet in Renal Disease Study equation
* Have a history or presence of medical illness including, but not limited to, any cardiovascular, thromboembolism or bleeding disorder, hepatic, respiratory, hematological, endocrine, immune, psychiatric or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study. In addition, participants with the following findings will be excluded: Confirmed Fridericia's corrected QT interval greater than (>)450 milliseconds (msec) for men and >470 msec for women. One additional ECG may be performed if required
* Have an elevated high-sensitivity C-reactive protein (>3 milligrams per Liter [mg/L]) or have a prothrombin time/international normalized ratio (PT/INR) or activated partial thromboplastin time (aPTT) >1.25 times (x) upper limit of normal (ULN)
* Are an investigator or site personnel directly affiliated or immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted
* Are Lilly employees or contractors or an immediate family member of such
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen
* Have donated more than 500 milliliters (mL) of blood within the past month
* Are unwilling to stop alcohol consumption while resident in the clinical research unit (CRU)
* Have an average weekly alcohol intake that exceeds 21 units per week (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Have an abnormal blood pressure (supine) defined as diastolic blood pressure >95 or less than (<)45 millimeters of Mercury (mmHg) and/or systolic blood pressure >160 or <90 mmHg. Re-testing may occur once during screening within 2 hours of the initial abnormal blood pressure measurement at the discretion of the investigator at screening
* Have positive findings for known drugs of abuse on urinary drug screening
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) virus nasopharyngeal polymerase chain reaction (PCR) test at Day -1
* Contact with SARS-CoV-2- positive or corona virus disease 2019 (COVID-19) patient within the last 14 days prior to admission to the clinical unit
* In the opinion of the investigator or the sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Day 137
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3473329 | Baseline up to Day 137
  PK: AUC of LY3473329
PK: Maximum Observed Drug Concentration (Cmax) of LY3473329 | Baseline up to Day 137
  PK: Cmax of LY3473329

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- [Derived] Nicholls SJ, Nissen SE, Fleming C, Urva S, Suico J, Berg PH, Linnebjerg H, Ruotolo G, Turner PK, Michael LF. Muvalaplin, an Oral Small Molecule Inhibitor of Lipoprotein(a) Formation: A Randomized Clinical Trial. JAMA. 2023 Sep 19;330(11):1042-1053. doi: 10.1001/jama.2023.16503. PMID 37638695